CLINICAL TRIAL: NCT00883155
Title: To Demonstrate the Relative Bioavailability of Bupropion HCI 100 mg Tablets Under Fasting Conditions.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B-09018
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2009-04

CONDITIONS: Healthy
Keywords: Antidepressant
MeSH Terms: interventions — Bupropion

ARMS (2):
- 1 (Experimental): Bupropion HCl 100 mg Tablets (Invamed Inc.)
  Interventions: Drug: Bupropion HCl 100 mg Tablets (Invamed Inc.)
- 2 (Active Comparator): Wellbutrin 100 mg Tablets (Glaxo Wellcome)
  Interventions: Drug: Wellbutrin 100 mg Tablets (Glaxo Wellcome)

INTERVENTIONS:
Drug: Bupropion HCl 100 mg Tablets (Invamed Inc.)
  Arms: 1
Drug: Wellbutrin 100 mg Tablets (Glaxo Wellcome)
  Arms: 2

SUMMARY:
To Demonstrate the Relative Bioavailability of Bupropion HCI 100 mg Tablets under Fasting Conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 1998-10; Primary Completion 1998-10 (Actual); Study Completion 1998-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Jameel Razack, M.D., Principal Investigator — Pharma Medica Research, Inc.